CLINICAL TRIAL: NCT05391269
Title: Histopathological Examination of Cases With Acute Appendicitis, A Retrospective Study at King Abdulaziz University Hospital, Jeddah, Saudi Arabia
Brief Title: Review of the Pathological Results of Appendectomy Specimens
Status: Completed | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dr. Mai Kadi, Assistant Professor, King Abdulaziz University
Other Study IDs: Histopathology of appendicitis
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Appendicitis; Pathology; Acute Appendicitis; Appendicitis (Diagnosis)
Keywords: Appendix; Pathology; Appendicitis diagnosis; Acute appendicitis
MeSH Terms: conditions — Appendicitis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective review study to evaluate the histopathological findings post appendectomy

DETAILED DESCRIPTION:
In this study, 940 cases will be reviewed. Patient demographics, accuracy of imaging modalities, and histopathological findings will be described.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent an appendectomy in king Abdulaziz university hospital in the period between 2010-2017

Exclusion Criteria:

* Any other patients will be excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent an appendectomy in king Abdulaziz university hospital in the period between 2010-2017
Sampling Method: Non-Probability Sample
Enrollment: 940 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Description of histopathological findings post appendectomy | 2010-2017
  Description of histopathological findings post appendectomy

SECONDARY OUTCOMES:
Relation between disease age, and gender | 2010-2017
  Relation between disease age, and gender
Assessment for accuracy of imagining modalities | 2010-2017
  Assessment for accuracy of imagining modalities

CONTACTS AND LOCATIONS:
Overall Officials: Mai S Kadi, MBBS, Principal Investigator — King Abdulaziz University, Jeddah, Saudi Arabia
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia